CLINICAL TRIAL: NCT07056517
Title: A Single-Dose, Open-label, Pharmacokinetics Study of Lobeglitazone From M107 ODT and Duvie® Under Fasted and Fed Conditions in Healthy Adults
Brief Title: Pharmacokinetics and Safety of M107 Orally Disintegrating Tablet in Healthy Adults
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Aclipse Two Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: M107-C101
Record Dates: First submitted 2025-06-30; First posted 2025-07-09 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-06

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- M107-C101 Cohort 1 (Experimental): Participants will receive a single oral dose of either Duvie (0.415 milligrams) or M107 Orally Disintegrating Tablet (0.4 milligrams) under fasted conditions on Day 1, followed by the alternate treatment on Day 8 after a 7-day washout. 8 participants are expected to enroll in this cohort.
  Interventions: Drug: M107 and Duvie - Cohort 1
- M107-C101 Cohort 2 (Experimental): Participants will receive a single 0.8 milligram oral dose of M107 Orally Disintegrating Tablet under fasted conditions on Day 1 and under fed conditions on Day 8, following a 7-day washout. 8 participants are expected to enroll in this cohort.
  Interventions: Drug: M107 - Cohort 2
- M107-C101 Cohort 3 (Experimental): Participants will receive a single 1.2 milligram dose of M107 Orally Disintegrating Tablet under fasted conditions. 8 participants are expected to enroll in this cohort.
  Interventions: Drug: M107 - Cohort 3

INTERVENTIONS:
Drug: M107 and Duvie - Cohort 1 — Dosage form - Oral tablets Dosage - Duvie 0.415 mg and M107 ODT 0.4 mg Participants will receive each treatment once under fasted conditions in a randomized two-period crossover design.
  Arms: M107-C101 Cohort 1
Drug: M107 - Cohort 2 — Dosage form - Orally disintegrating tablet Dosage - 0.8 mg Participants will receive M107 once under fasted conditions and once after a high-fat, high-calorie meal in a two-period crossover design.
  Arms: M107-C101 Cohort 2
Drug: M107 - Cohort 3 — Dosage form - Orally disintegrating tablet Dosage - 1.2 mg Participants will receive a single oral dose of M107 under fasted conditions.
  Arms: M107-C101 Cohort 3

SUMMARY:
Phase 1 study evaluating the safety, tolerability, and pharmacokinetics of lobeglitazone administered as M107 Orally Disintegrating Tablet and Duvie tablet in healthy adult participants under fasted and fed conditions.

DETAILED DESCRIPTION:
This is a Phase 1, single-center, parallel group study designed to determine the single-dose safety and PK profile of lobeglitazone from M107 ODT and Duvie, both administered orally in healthy adult volunteers.

Participants will be enrolled in 1 of 3 cohorts conducted in parallel:

Cohort 1 (Crossover): A single dose of Duvie oral tablet (0.415 mg; fasted) on Day 1 followed by a single dose of M107 ODT (0.4 mg; fasted) on Day 8, or vice versa, based on their random assignment with a 7-day washout between each dose.

Cohort 2 (Crossover): M107 ODT (0.8 mg; fasted) followed by M107 ODT (0.8 mg; fed) after a 7-day washout.

Cohort 3: M107 ODT (1.2 mg fasted) Participants in this cohort will receive M107 ODT 1.2 mg after a 10-hour fast.

A total of up to 24 participants are planned to be enrolled, 8 in each cohort, in order to ensure 6 evaluable participants in each cohort. At least 2 males and 2 females are to be enrolled in each cohort.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female participants aged 18 to 55 years (inclusive) at the time of informed consent.
2. Body Mass Index (BMI) between 18.0 and 30.0 kg/m² (inclusive) at Screening.
3. Body weight ≥50 kg at Screening.
4. Capable of giving informed consent and complying with study procedures.
5. Female participants must be of non-childbearing potential (postmenopausal or surgically sterile) or, if of childbearing potential, must agree to use acceptable contraception.
6. Participants must be non-smokers and must not have used any nicotine-containing products within 30 days prior to Screening and throughout the study.
7. Normal findings in physical examination, clinical laboratory tests, vital signs, and ECG, or findings considered not clinically significant by the investigator.
8. Willing to abstain from alcohol, grapefruit products, and caffeine as per study restrictions.
9. Willing to refrain from strenuous physical activity as specified in the protocol.
10. Male participants must agree to use contraception and avoid sperm donation during the study and for a specified period after.
11. Female participants of childbearing potential must agree to refrain from egg donation during the study and for at least 30 days after the last dose of study drug.

Exclusion Criteria:

1. Pregnant or breastfeeding females, or individuals (male or female) actively trying to conceive.
2. History of drug or alcohol use disorder within the past 2 years.
3. Active smoker or user of nicotine products (>5 cigarettes/week) or positive cotinine test at admission.
4. Difficulty with venipuncture or history of coagulopathy/endocarditis.
5. Significant history of cardiovascular, respiratory, gastrointestinal, renal, hepatic, neurological, endocrine, hematologic, or psychiatric disorders.
6. History of malignancy not in complete remission for at least 5 years (except localized basal/squamous cell skin cancer or prostate cancer deemed controlled).
7. Use of any prescription or over-the-counter medication, vitamins, or herbal supplements within 14 days or 5 half-lives prior to screening.
8. Use of any prescription medication, over-the-counter medication, or herbal supplements (other than permitted contraceptives or as approved by the investigator) from Screening until completion of the study.
9. Elevated resting blood pressure (systolic >140 mmHg or diastolic >90 mmHg) or heart rate >100 bpm.
10. History of major surgery within 4 weeks or minor surgery within 2 weeks of dosing.
11. Recent flu-like illness or respiratory infection within 2 weeks, or recent live-virus vaccination within 4 weeks of dosing.
12. Clinically significant ECG abnormalities including QTcF >450 ms, 2nd/3rd degree atrioventricular block, or incomplete left hemiblock.
13. Known bleeding disorders or history of significant allergic reaction to any drug component used in the study.
14. Blood or plasma donation >500 mL within 30 days before screening.
15. Any other condition which, in the opinion of the investigator, would preclude safe participation.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-07-11 (Actual); Primary Completion 2025-09-02 (Estimated); Study Completion 2025-09-02 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs), serious adverse events (SAEs), and clinically significant abnormalities | From screening to follow-up (up to Day 15 post-dose)
  To assess the frequency and severity of TEAEs, SAEs, and any clinically significant changes in laboratory parameters, vital signs, electrocardiogram, and physical examination findings following administration of M107 Orally Disintegrating Tablet and Duvie.
Maximum observed plasma concentration (Cmax) | From pre-dose to 48 hours post-dose
  To determine the peak plasma concentration of Lobeglitazone following oral administration of M107 Orally Disintegrating Tablet and Duvie.
Time to maximum observed plasma concentration (Tmax) | From pre-dose to 48 hours post-dose
  To assess the time it takes to reach the maximum plasma concentration of Lobeglitazone after administration.
Last measurable plasma concentration (Clast) | From pre-dose to 48 hours post-dose
  To evaluate the last quantifiable concentration of Lobeglitazone detected in plasma following administration.
Time of last measurable plasma concentration (Tlast) | From pre-dose to 48 hours post-dose
  To determine the time at which the last quantifiable plasma concentration of Lobeglitazone is observed.
Area under the concentration-time curve from 0 to 24 hours (AUC0-24h) | From pre-dose to 24 hours post-dose
  To evaluate the extent of Lobeglitazone exposure over the first 24 hours post-dose.
Area under the concentration-time curve from 0 to last measurable concentration (AUC0-last) | From pre-dose to 48 hours post-dose
  To assess the total plasma exposure to Lobeglitazone from dosing until the last quantifiable concentration.
Area under the concentration-time curve extrapolated to infinity (AUCinf) | From pre-dose to 48 hours post-dose
  To estimate total drug exposure by including the extrapolated portion of the concentration-time curve.
Percentage of AUC extrapolated (%AUCexp) | From pre-dose to 48 hours post-dose
  Percentage of the total area under the plasma concentration-time curve from time zero to infinity (AUC₀-inf) that is extrapolated beyond the last measurable concentration (%AUCexp).
Terminal elimination half-life (t½) | From pre-dose to 48 hours post-dose
  To determine the time required for the plasma concentration of Lobeglitazone to decrease by half during the terminal elimination phase.
Apparent oral clearance (CL/F) | From pre-dose to 48 hours post-dose
  To assess the rate at which Lobeglitazone is eliminated from the plasma after oral administration.
Apparent volume of distribution (Vz/F) | From pre-dose to 48 hours post-dose
  To calculate the apparent volume in which Lobeglitazone is distributed throughout the body after oral administration.
Terminal elimination rate constant (λz or Kel) | From pre-dose to 48 hours post-dose.
  To estimate the terminal elimination rate constant (λz or Kel) from the log-linear terminal phase of the plasma concentration-time curve following oral administration of lobeglitazone.

SECONDARY OUTCOMES:
Effect of food on maximum observed plasma concentration (Cmax) of Lobeglitazone | From pre-dose to 48 hours post-dose
  To compare the peak plasma concentration of Lobeglitazone after administration of M107 Orally Disintegrating Tablet under fasted versus fed conditions.
Effect of food on time to maximum observed plasma concentration (Tmax) of Lobeglitazone | From pre-dose to 48 hours post-dose
  To assess the difference in time to reach peak plasma concentration under fasted versus fed conditions following administration of M107 Orally Disintegrating Tablet.
Effect of food on total drug exposure (AUC0-last and AUCinf) | From pre-dose to 48 hours post-dose
  To evaluate the area under the concentration-time curve from time zero to last measurable concentration (AUC0-last) and extrapolated to infinity (AUCinf) for Lobeglitazone under fasted versus fed conditions.
Effect of food on terminal elimination half-life (t½) | From pre-dose to 48 hours post-dose
  To compare the terminal elimination half-life of Lobeglitazone under fasted and fed conditions following administration of M107 Orally Disintegrating Tablet.
Effect of food on apparent oral clearance (CL/F) and volume of distribution (Vz/F) | From pre-dose to 48 hours post-dose
  To evaluate differences in oral clearance and volume of distribution of Lobeglitazone when M107 Orally Disintegrating Tablet is administered under fed versus fasted conditions.
Effect of food on terminal elimination rate constant (λz or Kel) of lobeglitazone | From pre-dose to 48 hours post-dose.
  To compare the terminal elimination rate constant (λz or Kel) of lobeglitazone under fasted and fed conditions following administration of the M107 Orally Disintegrating Tablet.

CONTACTS AND LOCATIONS:
Locations (1):
- Nucleus Network Pty Ltd., Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No